CLINICAL TRIAL: NCT07129291
Title: Development of Dual Language (Urdu and English) Digital Software For Self- Assessment And Management Of Adult Dysarthria Patients
Brief Title: Development of Dual Language (Urdu and English) Digital Software for SA, Management Of Adult Dysarthria
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PhDRSW/Batch-Fall23/2226
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Dysarthria
MeSH Terms: conditions — Dysarthria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dual-Language Dysarthria Self-Assessment and Management Software (D-SAMS) (Experimental): D-SAMS is a bilingual (Urdu and English) digital tool designed for adult dysarthria patients. It enables users to assess their speech through interactive tasks (e.g., repetition, reading, and pronunciation exercises), receive feedback, and track progress over time. The software includes audio-visual prompts, self-rating scales, and progress charts, and is tailored to accommodate varying levels of dysarthria severity. It supports independent practice and helps speech-language pathologists monitor patients remotely
  Interventions: Combination Product: Experimental: Dual-Language Dysarthria Self-Assessment and Management Software (D-SAMS)

INTERVENTIONS:
Combination Product: Experimental: Dual-Language Dysarthria Self-Assessment and Management Software (D-SAMS) — D-SAMS is a bilingual (Urdu and English) digital tool designed for adult dysarthria patients. It enables users to assess their speech through interactive tasks (e.g., repetition, reading, and pronunciation exercises), receive feedback, and track progress over time. The software includes audio-visual prompts, self-rating scales, and progress charts, and is tailored to accommodate varying levels of dysarthria severity. It supports independent practice and helps speech-language pathologists monitor patients remotely

SUMMARY:
The research focuses on the development of a dual-language (Urdu and English) digital software designed for the self-assessment and management of adult dysarthria patients. Dysarthria, a motor speech disorder resulting from neurological injury, significantly affects an individual's ability to communicate effectively.

DETAILED DESCRIPTION:
Current assessment tools are often clinician-dependent and predominantly available in English, limiting accessibility for non-English speakers, especially in Pakistan and other Urdu-speaking regions. This study aims to bridge that gap by creating a user-friendly, culturally relevant, and linguistically accessible software platform. The software will enable adult dysarthric patients to monitor their speech abilities, track progress, and participate more actively in their therapy process. It is expected to enhance patient autonomy, improve communication outcomes, and support speech-language pathologists in delivering more efficient care. The dual-language interface ensures broader usability, promoting inclusion and better engagement among diverse user groups in bilingual settings.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18+) diagnosed with dysarthria due to neurological causes (e.g., stroke, Parkinson's).
* Able to understand and communicate in Urdu and/or English.
* Cognitive ability sufficient to use digital tools for self-assessment.
* Consent to participate in the study.

Exclusion Criteria:

* Severe cognitive impairment or dementia limiting participation.
* Co-existing speech disorders unrelated to dysarthria (e.g., aphasia).
* Hearing impairments that prevent use of audio-based software.
* Unwillingness or inability to use digital devices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2025-04-17 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Frenchay Dysarthria Assessment (FDA-2) | 24 Months
  Assesses: Motor speech function. Scoring: A (normal) to E (severely impaired) across speech subsystems.
Dysarthria Impact Profile (DIP) | 24 Months
  Assesses: Psychosocial impact of dysarthria. Scoring: 48 items, rated 1-5; higher scores = greater negative impact.
Speech Intelligibility Rating Scale (SIRS) | 24 Months
  Assesses: Speech clarity. Scoring: 1 (unintelligible) to 5 (fully intelligible).
Voice Handicap Index-10 (VHI-10) (optional) | 24 Months
  Assesses: Patient's perception of voice issues. Scoring: 0-4 per item; total out of 40. Higher = more voice difficulty.

CONTACTS AND LOCATIONS:
Locations (1):
- Rehabilitation Centers in Punjab, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No